CLINICAL TRIAL: NCT04384718
Title: Assessing the Generalizability of the Tachidino Protocol for Intervention on Reading and Spelling Disorders to Different Clinical Contexts
Brief Title: Assessing the Generalizability of the Tachidino Protocol to Different Clinical Contexts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: University of Urbino "Carlo Bo" (Other); Asur Marche - AV1 - Centre for Clinical Child Neuropsychology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 05-20 oss (to be confirmed)
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Developmental Dyslexia
Keywords: Developmental Dyslexia; Intervention; Hemisphere-specific stimulation; Visual-attentional training; telerehabilitation
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Medea Group: Group of children with Developmental Dyslexia treated with Tachidino protocol at IRCCS Medea
- Asur Group: Group of children with Developmental Dyslexia treated with Tachidino protocol at Asur Marche
- Waiting list Group: Group of children with Developmental Dyslexia on a waiting list for treatment with Tachidino protocol at IRCCS Medea or Asur Marche

SUMMARY:
The study aims to document the effectiveness and acceptability of the intervention system for specific reading and writing disorders, in use at Scientific Institute (IRCCS) Medea, as applied and adapted to a different clinical context and socio-demographic situation. To this purpose, two groups of children will be recruited and treated in two different contexts, and treatment outcomes will be compared. The first one is the centre where the Tachidino platform has been developed and validated, the second one is a different centre, in a different geographical region where lower digital alphabetization may be a disadvantaging factor, but lower population density and the presence of fewer centres for assessment and intervention for learning disorders make remotely monitored protocols even more valuable.

DETAILED DESCRIPTION:
Specifically, the intervention system based on the web platform "Tachidino" and routinely used for the rehabilitation of reading and spelling disorders at Medea, Lombardy region, would be extended to Marche (precisely, the clinical service connected to Urbino University, located in Pesaro, a coastal town in Central Italy), a different geographical region with different population characteristics. Precisely, the Lombardy region is a highly industrialized region with the highest digitalization rate in Italy, whereas Marche is a more agriculture-oriented region, with lower population density and less widespread use of digital technologies. The main aim of the study is, then, to ascertain whether the effectiveness levels found for the treatment protocol in the original context generalize to a different context and population.

The system for the empowerment of reading and spelling skills ("Tachidino" software) is based on two principles of proven effectiveness:

1. The selective stimulation of a cerebral hemisphere and specific reading strategies.
2. The training of selective visuospatial attention, as well as the perception of rapid movement and the control of visual crowding effects.

Clinical and assessment procedures

In current clinical practice at IRCCS Medea, intervention in "e-health" mode is divided into one or more rehabilitation modules through the use of the Tachidino platform, with systematic monitoring and motivational reinforcement by professionals with experience in e-health approaches. In order to be included in the training, the child must have already obtained a diagnosis of dyslexia, according to the current diagnostic standards.

The structure of the intervention modules is as follows:

* 1 initial meeting to get to know the child, pre-test assessment - reading and writing tests of words, non-words and sentences, metaphonological tests and text reading tests (reading accuracy and speed) in order to define dyslexia subtypes; intervention planning - demonstration of Tachidino use and programming of first activities
* telephone support to monitor and motivate correct use of the software, during active intervention
* 1 final assessment meeting (with repetition of the tests used at pre-test and compilation of questionnaires).

In addition to the main goal and the above-described procedure, the study will investigate the effects of treatment with additional tests providing parallel versions and lists of stimuli, so as to exclude any possible repetition effect and thus to better highlight "pure" intervention effects.

Participants' characteristics: Children aged between 7 and 16 years with a diagnosis of Specific Reading Disorder, Mixed Disorder of Scholastic Skills or Developmental Dyslexia, pertaining to International Classification of Diseases (ICD-10) codes F81, F81.0, F81.3, referred to one of the two participating centres because of school learning problems.

Total number of subjects: 32 (16 per centre). An additional group of 16 children with Dyslexia and/or Dysgraphia on a waiting list will also be tested and retested after 4 weeks, providing a further control for the effects of intervention.

The number of participants has been determined with a power analysis based on data on the effects of treatment observed in the group already treated with Tachidino at IRCCS Medea. The number of 32 participants turned out to be sufficient to provide a power of 0.8 with alpha set at .005.

ELIGIBILITY:
Inclusion Criteria:

* A formal diagnosis of Developmental Dyslexia, Specific Reading Disorders, or Mixed Scholastic Learning Disorders
* Age between 7 and 16
* Attending at least the third class of primary school
* Monolingual speakers of Italian or bilingual speakers with perfect mastery of the Italian language (equivalent to monolinguals)
* Intelligence Quotient (IQ) >= 80
* At least one z-score below -2 Standard Deviations from age mean in at least one of the following tests: text reading, word reading, nonword reading ("DDE-2" battery, "MT" tests)
* Not having received any specific rehabilitation treatment for dyslexia before

Exclusion Criteria:

* Intellectual disability
* Neurological disorders
* Sensory deficits that are not /cannot be corrected-to-normal by lenses or hearing aids.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be recruited among those referred to either IRCCS Medea or ASUR Marche because of learning and school-achievement problems. All children who were offered treatment through the web-based platform "Tachidino" and who meet inclusion/ exclusion criteria will be enrolled in the study after their parents have accepted and signed informed consent. After completion of the two treatment groups (32 children), the next 16 children referred to either Centre will be enrolled as Waiting list group and treated after a 4 weeks observation period without treatment.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
change from pre-test to post-test in reading ability | 4 weeks
  Difference in treatment-related changes (post-test minus pre-test) observed in reading measures (speed and accuracy in word, nonword and text reading standardized tests: Memory Training (MT) group reading test and "Developmental Dyslexia and Dysgraphia" (DDE-2); average of the scores expressed as z-scores with respect to age norms)

SECONDARY OUTCOMES:
change from pre-test to post-test in metaphonological ability | 4 weeks
  Difference in treatment-related changes (post-test minus pre-test) observed in metaphonological tests (phonemic analysis and phoneme blending) - average of the number of errors in the two tests
change from pre-test to post-test in short-term-memory | 4 weeks
  Difference in treatment-related changes (post-test minus pre-test) observed in memory tests (direct and indirect span) - average of the number of correct responses in the two tests
change from pre-test to post-test in executive functions | 4 weeks
  Difference in treatment-related changes (post-test minus pre-test) observed in executive functions tests (go-no-go paradigm) - average of the number of correct responses in the two tests
difference in change between treated and untreated children | 4 weeks
  Difference found in pre-post test changes (post-test minus pre-test) observed in reading tests (reading speed and accuracy measured with "MT tests" and "DDE-2") - expressed as z-scores according to age, between the two groups treated with Tachidino remotely delivered intervention and the waiting list group

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Lorusso, Ph.D., Principal Investigator — IRCCS E. Medea
Locations (3):
- Italy (3):
  - Scientific Institute IRCCS E. Medea, Bosisio Parini, LC
  - ASUR Marche, Centre for Clinical Child Neuropsychology, Pesaro
  - University of Urbino, Urbino